CLINICAL TRIAL: NCT05353764
Title: Effect of Scalp Nerve Block Combined With Intercostal Nerve Block on Quality of Recovery After Deep Brain Stimulation in Patients With Parkinson's Disease
Brief Title: Effect of Scalp Nerve Block on the Recovery Quality of Parkinson's Patients After Deep Brain Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Wen-bin Lu, MD, Attending doctor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SNB-QoR
Record Dates: First submitted 2022-04-19; First posted 2022-04-29 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SNB group (Experimental): patients in the SNB group will receive general anesthesia combined with scalp nerve block and intercostal nerve block with 0.5% ropivacaine.
  Interventions: Other: scalp nerve block combined with intercostal nerve block using 0.5% ropivacaine
- control group (No Intervention): patients in control group will receive general anesthesia without nerve block.

INTERVENTIONS:
Other: scalp nerve block combined with intercostal nerve block using 0.5% ropivacaine — Participants randomized to the SNB group will receive general anesthesia combined with scalp nerve block and intercostal nerve block with 0.5% ropivacaine, which was performed exclusively by an attending anesthesiologist.An attending anesthesiologist will select the site of SNB based on the surgical incision site. Scalp nerve was blocked including greater occipital nerve (2-3ml), superficial temporal nerve (2-3ml), trochlear nerve (2-3ml) and supraorbital nerve (2-3ml). The total volume in scalp nerve block will not exceed 10 ml.Ultrasound-guided unilateral ICNB will be performed at the level of T4-T5 next to the sternum.10-15ml of 0.5% ropivacaine will be injected into the intercostal spaces where incision locates after negative aspiration.
  Arms: SNB group

SUMMARY:
Patients diagnosed with Parkinson's disease (PD) undergoing deep Brain Stimulation (DBS) have a higher risk of perioperative complications and postoperative pain will affect quality of recovery (QoR) resulting in longer hospitalization time and higher hospital costs. Scalp nerve block (SNB) combined with intercostal nerve block (ICNB)can alleviate postoperative pain while effect of them on postoperative recovery quality of patients diagnosed with PD was unclear. Therefore, the investigators conducted a randomized controlled trails to provide a novel method for enhanced recovery and early prevention and treatment of acute pain after DBS surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients with PD who receive elective deep brain stimulation (DBS) surgery
* Aged ≥ 18
* American Society of Anesthesiologists (ASA) physical status of I-III
* Able to communicate normally

Exclusion Criteria:

* Allergy to local anesthetics
* Pre-existing infection at block site
* Severe coagulopathy
* Pre-existing neuropathic pain condition
* Previous history of DBS surgery
* unwilling to provide informed consent or poor compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
The 15-item QoR score | 24 hour after surgery
  The 15-item QoR score is used to asses quality of recovery after surgery which ranges 0-150 and higher QoR-15 scores indicate better postoperative recovery

SECONDARY OUTCOMES:
The 15-item QoR score | 72 hour and 1 month after surgery
  The 15-item QoR score is used to asses quality of recovery after surgery which ranges 0-150 and higher QoR-15 scores indicate better postoperative recovery
The NRS score | before discharge from PACU, at 24 hour, 72 hour and 1 month after surgery
  Postoperative pain will be quantified using the NRS ranging from 0 to 10, where 0 means "no pain at all" and 10 means "the worst pain imaginable"
The patients with PONV | 24 hour after surgery
  postoperative nausea and vomiting
Consumption of opioid | during operation
  The consumption of opioid reffers to remifentanil consumption

CONTACTS AND LOCATIONS:
Overall Officials: Xiya Yu, M.D, Principal Investigator — Changhai hospital, Shanghai, China
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Sheng Y, Wang H, Chang X, Jin P, Lin S, Qian S, Xie J, Lu W, Yu X. Effect of Scalp Nerve Block Combined with Intercostal Nerve Block on the Quality of Recovery in Patients with Parkinson's Disease after Deep Brain Stimulation: Protocol for a Randomized Controlled Trial. Brain Sci. 2022 Jul 29;12(8):1007. doi: 10.3390/brainsci12081007. PMID 36009070